CLINICAL TRIAL: NCT01757366
Title: Safety and Efficacy of Ginsenoside Rg3 in Combination With First-line Chemotherapy in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBTH102
Record Dates: First submitted 2012-12-21; First posted 2012-12-28 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2012-12

CONDITIONS: Self Efficacy
MeSH Terms: interventions — ginsenoside Rg3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): Ginsenoside Rg3 plus First-line Chemotherapy
  Interventions: Drug: Ginsenoside Rg3 plus First-line Chemotherapy
- Active Comparator (Active Comparator): First-line Chemotherapy
  Interventions: Drug: First-line Chemotherapy

INTERVENTIONS:
Drug: Ginsenoside Rg3 plus First-line Chemotherapy — Ginsenoside Rg3 20mg 2/day po,patients will receive Ginsenoside Rg3 until progression
  XELOX(oxaliplatin 130mg/m2 iv d1;capecitabine 1000mg/m2 po bid d1-14)every 3 weeks for 4 cycles followed by capecitabine until progression
  Arms: experimental
Drug: First-line Chemotherapy — XELOX(oxaliplatin 130mg/m2 iv d1;capecitabine 1000mg/m2 po bid d1-14)every 3 weeks for 4 cycles followed by capecitabine until progression
  Arms: Active Comparator

SUMMARY:
Safety and Efficacy of Ginsenoside Rg3 in Combination with First-line Chemotherapy in Advanced Gastric Cancer.The purpose of this study is to assess the safety of Ginsenoside Rg3 in advanced gastric cancer, and whether it improves the efficacy of first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1;
3. Histologically or cytologically confirmed gastric cancer;
4. At least have one measurable disease(according to RECIST, Response Evaluation Criteria in Solid Tumors )
5. Life expectancy of at least 3 months;

Exclusion Criteria:

1. Received any prior treatment including Ginsenoside Rg3;
2. Active or uncontrolled infection;
3. Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
4. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
Overall Survival (OS) | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liu, Principal Investigator — Hebei Tumor Hospital
Locations (1):
- Hebei Tumor Hospital, Shijiazhuang, Hebei, China